CLINICAL TRIAL: NCT07110571
Title: A Multi-cohort, Multi-center Phase II Clinical Study of Adebrelimab in Combination With SHR-A1811/SHR-A1904 and Chemotherapy or Adebrelimab in Combination With SHR-8068 as the Treatment in Subjects With Gastric or Gastroesophageal Junction Cancer
Brief Title: A Trial of Adebrelimab Plus (SHR-A1811/SHR-A1904 With Chemotherapy) or SHR-8068 as Treatment for Gastric/GEJ Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316-205
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Gastric Cancer; Gastroesophageal-junction Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A - Adebrelimab in combination with SHR-A1811 and chemotherapy (Experimental)
  Interventions: Drug: Adebrelimab Injection; Drug: SHR-A1811 for Injection
- Cohort B - Adebrelimab in combination with SHR-A1904 (Experimental)
  Interventions: Drug: Adebrelimab Injection; Drug: SHR-A1904 for Injection
- Cohort D - Adebrelimab in combination with SHR-8068 (Experimental)
  Interventions: Drug: Adebrelimab Injection; Drug: SHR-8068 Injection

INTERVENTIONS:
Drug: Adebrelimab Injection — Adebrelimab injection.
Drug: SHR-A1811 for Injection — SHR-A1811 for injection.
  Arms: Cohort A - Adebrelimab in combination with SHR-A1811 and chemotherapy
Drug: SHR-A1904 for Injection — SHR-A1904 for injection.
  Arms: Cohort B - Adebrelimab in combination with SHR-A1904
Drug: SHR-8068 Injection — SHR-8068 injection.
  Arms: Cohort D - Adebrelimab in combination with SHR-8068

SUMMARY:
This is a multi-cohort, multi-center Phase II clinical study exploring the efficacy of treatment with either Adebrelimab plus SHR-A1811/SHR-A1904 and chemotherapy, or Adebrelimab plus SHR-8068 in patients with gastric or gastroesophageal junction (GEJ) cancer. The study also evaluates the safety and tolerability of these combination regimens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed gastric or gastroesophageal junction adenocarcinoma who have not received prior anti-tumor therapy for gastric/gastroesophageal junction cancer.
2. Age: ≥18 and ≤70 years, both male and female.
3. Ability to provide fresh tumor tissue (preferred) or archival formalin-fixed paraffin-embedded (FFPE) tumor blocks/unstained slides obtained within 6 months before enrollment.
4. Availability of biomarker testing results before enrollment.
5. ECOG performance status of 0-1.
6. Life expectancy ≥ 6 months.
7. Adequate organ and bone marrow function.
8. Female participants must be either non-childbearing potential or of childbearing potential with a negative serum pregnancy test within 3 days prior to treatment initiation and not lactating. Childbearing-potential participants and their partners must agree to avoid sperm/ovum donation and comply with contraception requirements from informed consent signing until 8 months after the last dose.
9. Voluntarily signed informed consent form, with willingness and ability to comply with scheduled visits, treatments, laboratory tests, and study procedures.

Exclusion Criteria:

1. Known squamous cell carcinoma, undifferentiated carcinoma, mixed adenocarcinoma with other histologic types, or other non-adenocarcinoma gastric cancers.
2. 20% body weight loss within 2 months before enrollment.
3. Prior treatments: Anti-tumor therapy for gastric/gastroesophageal junction cancer; Participation in other drug trials with last dose ≤4 weeks or ≤5 half-lives (whichever longer) before enrollment; Major surgery within 28 days before enrollment; Live attenuated vaccination within 28 days before enrollment or planned during/within 60 days after treatment.
4. Known hypersensitivity to any study drug component (Adebrelimab, SHR-A1811, SHR-A1904, SHR-8068, fluorouracil, capecitabine, tegafur/gimeracil/oteracil) or humanized monoclonal antibodies.
5. Other malignancies within 5 years, except curatively treated basal/squamous cell skin cancer, superficial bladder cancer, cervical carcinoma in situ, ductal breast carcinoma in situ, or papillary thyroid cancer.
6. History of immunodeficiency, organ transplantation, or active autoimmune disease.
7. Clinically significant bleeding within 3 months or bleeding predisposition at screening; Arterial/venous thromboembolism within 6 months or at screening.
8. Non-healing wounds, active ulcers, or untreated fractures.
9. Active severe gastrointestinal disorders.
10. Interstitial pneumonia or lung disease.
11. Severe cardiovascular/cerebrovascular diseases or metabolic disorders.
12. Active HBV/HCV infection or HBV-HCV co-infection.
13. Active tuberculosis (TB) within 1 year by history/CT, or prior untreated active TB >1 year ago.
14. Severe infection within 4 weeks before first dose; CTCAE ≥Grade 2 active infection requiring systemic antibiotics within 2 weeks; Chronic infections potentially affecting treatment/surgery.
15. History of drug abuse or illicit substance use.
16. Other conditions that may increase study risk, confound results, or render the patient unsuitable per investigator judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate assessed by the Pathology Review Committee (PRC). | Approximately 13 weeks.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) evaluated per NCI-CTCAE v5.0. | Approximately 1 year.
Incidence and severity of serious adverse events (SAEs) evaluated per NCI-CTCAE v5.0. | Approximately 1 year.
Major pathological response (MPR) rate assessed by the Pathology Review Committee (PRC). | Approximately 13 weeks.
Pathological complete response (pCR) rate evaluated by the investigational site's pathology assessment. | Approximately 13 weeks.
Event-Free Survival (EFS). | Approximately 1 year.
Disease-Free Survival (DFS). | Approximately 1 year.
Objective Response Rate (ORR). | Approximately 1 year.
Overall Survival (OS). | Approximately 2 years.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided